CLINICAL TRIAL: NCT00267319
Title: Fatigue Outcomes of Copaxone Users in Relapsing-remitting Multiple Sclerosis
Brief Title: FOCUS Fatigue Outcome in Copaxone USers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR4002A_4002
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

ARMS (1):
- single group (Experimental)
  Interventions: Drug: Glatiramer acetate

INTERVENTIONS:
Drug: Glatiramer acetate

SUMMARY:
* The study primarily investigates the effect of copaxone on fatigue during treatment, compared to baseline in patients with relapsing-remitting multiple sclerosis.
* Secondary outcome measures are:disability, relapse rate, quality of life and depression.

ELIGIBILITY:
Inclusion Criteria:

* relapsing-remitting Multiple Sclerosis (MS),
* at least 2 relapses in previous 2 years prior to copaxone or interferon beta treatment,
* ambulant patients i.e disability score EDSS MAX 5,5,
* clinically stable MS
* relapse free and steroid free at least 30 days prior to start copaxone treatment

Exclusion Criteria:

* hypersensitivity to glatiramer acetate or mannitol,
* pregnancy,
* fertile female not willing to use effective contraception,
* previous treatment with copaxone

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
fatigue impact scale | at baseline, month 6 and month 12

SECONDARY OUTCOMES:
relapse rate | at baseline, month 6 and month 12
quality of life | at baseline, month 6 and month 12
depression | at baseline, month 6 and month 12
disability | at baseline, month 6 and month 12
Adverse events | at baseline, month 6 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Priborska, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Prague, Czechia